CLINICAL TRIAL: NCT00920088
Title: A Phase I Study to Evaluate the Effect of Darunavir/Ritonavir and Lopinavir/Ritonavir on GSK2248761 Pharmacokinetics and to Assess the Effect of GSK2248761 on CYP450 Probe Drugs in Healthy Adult Subjects
Brief Title: Drug Interaction Study of Darunavir/Ritonavir and Lopinavir/Ritonavir on GSK2248761 PK and CYP450 Probe Drugs
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: E.D. Derilus; Clinical Disclosure Advisor, GSK Clinical Disclosure
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 113045
Record Dates: First submitted 2009-06-12; First posted 2009-06-15 (Estimated); Last update posted 2010-11-03 (Estimated); Status verified 2010-11

CONDITIONS: Healthy Subjects; Infection, Human Immunodeficiency Virus
Keywords: probes; NNRTI; drug interaction; protease inhitibor
MeSH Terms: conditions — Infections; Acquired Immunodeficiency Syndrome | interventions — Darunavir; Ritonavir; Lopinavir; Midazolam; Dextromethorphan; Flurbiprofen; IDX 899

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): GSK2248761 with LPV/RTV arm and probes
  Interventions: Drug: lopinavir/ritonavir; Drug: Midazolam; Drug: Dextromethorphan; Drug: Flurbiprofen; Drug: GSK2248761
- Cohort 2 (Experimental): GSK2248761 with DRV/RTV
  Interventions: Drug: darunavir/ritonavir; Drug: GSK2248761

INTERVENTIONS:
Drug: darunavir/ritonavir — DRV/RTV 600/100mg
  Arms: Cohort 2
Drug: lopinavir/ritonavir — LPV/RTV 400/100mg
  Arms: Cohort 1
Drug: Midazolam — Midazolam 3mg
  Arms: Cohort 1
Drug: Dextromethorphan — Dextromethorphan 30mg
  Arms: Cohort 1
Drug: Flurbiprofen — Flurbiprofen 50mg
  Arms: Cohort 1
Drug: GSK2248761 — NNRTI under investigation

SUMMARY:
The purpose of this study is to evaluate the effect of GSK2448761 on CYP450 metabolic probes and to evaluate the 2-way interaction between GSK2448761 and two ritonavir-boosted protease inhibitors that are commonly used in HIV-infected subjects.

ELIGIBILITY:
Inclusion Criteria:

* Healthy as determined by a responsible and experienced physician, based on a medical evaluation including medical history, physical examination, laboratory tests and cardiac monitoring.
* Male or female between 18 and 50 years of age inclusive, at the time of signing the informed consent.
* A female subject is eligible to participate if she is of non-childbearing potential (i.e., physiologically incapable of becoming pregnant).
* Male subjects must agree to use one of the contraception methods listed in the protocol. This criterion must be followed from the time of the first dose of study medication until the follow-up visit.
* Body weight >=50 kg for men and >=45 kg for women and body mass index (BMI) within the range 18.5-31.0 kg/m2 (inclusive).
* Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the consent form.

Exclusion Criteria:

* As a result of the medical interview, physical examination, or screening investigations, the Investigator considers the subject unfit for the study.
* The subject has a positive pre-study drug/alcohol screen.
* Unwilling to refrain from the use of illicit drugs and adhere to other protocol-stated restrictions while participating in the study.
* History of regular alcohol consumption within 6 months of the study.
* Unwilling to abstain from alcohol for 48 hours prior to the start of dosing until collection of the final pharmacokinetic sample during each treatment period.
* History or regular use of tobacco- or nicotine-containing products within 3 months prior to screening.
* History/evidence of symptomatic arrhythmia, angina/ischemia, coronary artery bypass grafting (CABG) surgery or percutaneous transluminal coronary angioplasty (PCTA) or any clinically significant cardiac disease.
* History/evidence of clinically significant pulmonary disease.
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
* Subjects with a pre-existing condition interfering with normal gastrointestinal anatomy or motility, hepatic and/or renal function, that could interfere with the absorption, metabolism, and/or excretion of the study drugs. Subjects with a history of cholecystectomy should be excluded.
* The subject has participated in a clinical trial and has received an investigational product within the following time period prior to the first dosing day in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
* The subject has received GSK2248761 in a previous clinical trial.
* Use of prescription or non-prescription drugs, including vitamins, herbal and dietary supplements (including St John's Wort) within 7 days (or 14 days if the drug is a potential enzyme inducer) or 5 half-lives (whichever is longer) prior to the first dose of study medication, unless in the opinion of the Investigator and GSK Medical Monitor the medication will not interfere with the study procedures or compromise subject safety.
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation.
* Where participation in the study would result in donation of blood or blood products in excess of 500 mL within a 56 day period.
* Has a known intolerance or hypersensitivity to aspirin, NSAIDS, or benzodiazepines, or a known intolerance to the active and/or inactive ingredients in dextromethorphan, midazolam and flurbiprofen (Cohort 1 only)
* Has any condition or symptom contraindicated for administration of the study drugs: dextromethorphan, midazolam and flurbiprofen. The Investigator should reference the product information of each study drug. (Cohort 1 only)
* History of sensitivity to heparin or heparin-induced thrombocytopenia (if heparin is used to maintain the patency of an intravenous cannula).
* A positive pre-study Hepatitis B surface antigen or positive Hepatitis C antibody result within 3 months of screening.
* A positive test for HIV antibody.
* AST, ALT, alkaline phosphatase and bilirubin >=1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
* Pregnant females as determined by positive serum hCG test at screening or prior to dosing.
* Lactating females.
* The subject's systolic blood pressure is outside the range of 90-140mmHg, or diastolic blood pressure is outside the range of 45-90mmHg or heart rate is outside the range of 50-100bpm for female subjects or 45-100 bpm for male subjects at Screening and Day -1.
* Cardiac conduction abnormalities denoted on a single 12-lead ECG at screening or Day -1

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2009-06; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
PK parameters | 35 days

SECONDARY OUTCOMES:
12-lead ECGs | 35 days
clinical laboratory assessments | 35 days
vital signs | 35 days
pharmacokinetic parameters | 35 days

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (1):
- GSK Investigational Site, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Piscitelli S, Kim J, Gould E, Lou Y, White S, de Serres M, Johnson M, Zhou XJ, Pietropaolo K, Mayers D. Drug interaction profile for GSK2248761, a next generation non-nucleoside reverse transcriptase inhibitor. Br J Clin Pharmacol. 2012 Aug;74(2):336-45. doi: 10.1111/j.1365-2125.2012.04194.x. PMID 22288567